CLINICAL TRIAL: NCT05447897
Title: A Systematic Approach to Designing an Implementation Strategy to Increase Lung Cancer Screening and Smoking Cessation Treatment Among Federally Qualified Community Health Center Patients Who Smoke
Brief Title: Designing an Implementation Strategy for Lung Screening and Smoking Cessation Treatment in Community Health Centers
Acronym: SAILS-FQHC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22-215; P50CA244433-03S3 (NIH)
Record Dates: First submitted 2022-06-29; First posted 2022-07-07 (Actual); Results first posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-03

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stakeholder Advisory Group (Other): To co-design an implementation strategy that targets critical components in the delivery of SCT or LCS services for patients who smoke.
  Convene a stakeholder advisory group (CHC providers, quality improvement specialists, community engagement staff, and specialty providers) to review the results of the literature review and quantitative analysis of deidentified data in order to select a set of implementation strategies from a menu of strategies to implement. The team will meet with the stakeholder advisory group four times for 1-2 hours each.
  Interventions: Other: Qualitative Group Interviews; Other: Stakeholder advisory group

INTERVENTIONS:
Other: Qualitative Group Interviews — One time interview, 60-90 minutes
Other: Stakeholder advisory group — The team will meet with the stakeholder advisory group four times for 1-2 hours each

SUMMARY:
Tobacco use is the leading preventable cause of death in the US and a major driver of health disparities. Among our tools for reducing the harms of tobacco is lung cancer screening (LCS). This study will combine a review of existing qualitative and quantitative data on barriers to lung cancer screening and smoking cessation in underserved populations, a quantitative analysis of predictors of lung cancer screening and smoking cessation treatment use among Massachusetts Federally Qualified Health Centers (FQHC)s, and a stakeholder advisory group to synthesize these data and select implementation strategies that reflects the critical determinants and the strengths and resource constraints of the Federally Qualified Health Centers (FQHC) context.

DETAILED DESCRIPTION:
Aim 1) To design an implementation strategy that targets critical components in the delivery of SCT or LCS services for patients who smoke.

Aim 2) To assess the acceptability, appropriateness and feasibility of the implementation strategy among community health center staff.

ELIGIBILITY:
Inclusion Criteria:

FQHC implementation team including staff in the intervention FQHCs and their lung screening partners

Exclusion Criteria:

FQHC staff or partners who leave the organization before end of study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gina Kruse, MD, MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- Massacusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation

RESULTS

PARTICIPANT FLOW:
Groups:
- Stakeholder Advisory Group: To co-design an implementation strategy that targets critical components in the delivery of SCT or LCS services for patients who smoke.
  Convene a stakeholder advisory group (CHC providers, quality improvement specialists, community engagement staff, and specialty providers) to review the results of the literature review and quantitative analysis of deidentified data in order to select a set of implementation strategies from a menu of strategies to implement. The team will meet with the stakeholder advisory group four times for 1-2 hours each.
  Qualitative Group Interviews: One time interview, 60-90 minutes
  Stakeholder advisory group: The team will meet with the stakeholder advisory group five to six times for 0.5-1 hours each
Period: Overall Study
Arm/Group | Stakeholder Advisory Group
Started | 9
Completed | 7
Not Completed | 2
Not completed — Did not participate in survey | 2

BASELINE CHARACTERISTICS:
Groups:
- Stakeholder Advisory Group: To co-design an implementation strategy that targets critical components in the delivery of SCT or LCS services for patients who smoke.
  Convene a stakeholder advisory group (CHC providers, quality improvement specialists, community engagement staff, and specialty providers) to review the results of the literature review and quantitative analysis of deidentified data in order to select a set of implementation strategies from a menu of strategies to implement. The team will meet with the stakeholder advisory group five to six times for 0.5-1 hours each.
  Qualitative Group Interviews: One time interview, 60-90 minutes
  Stakeholder advisory group: The team will meet with the stakeholder advisory group five to six times for 0.5-1 hours each
Arm/Group | Stakeholder Advisory Group
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Intervention Measure
Description: Feasibility of Intervention Measure, 5-point Likert scales (range 1-5), higher values reflect favorable outcomes
Time Frame: End of study, up to 16 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Stakeholder Advisory Group
Number analyzed (Participants) | 7
units on a scale | 4 [3.25 to 5]

2. Secondary Outcome: Acceptability of Intervention Measure
Description: Acceptability of Intervention Measure, 5-point Likert scales (range 1-5), higher values reflect favorable outcomes
Time Frame: End of study, up to 16 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Stakeholder Advisory Group
Number analyzed (Participants) | 7
units on a scale | 4 [4 to 5]

3. Secondary Outcome: Intervention Appropriateness Measure
Description: Intervention appropriateness measure, 5-point Likert scales (range 1-5), higher values reflect favorable outcomes
Time Frame: End of study, up to 16 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Stakeholder Advisory Group
Number analyzed (Participants) | 7
units on a scale | 4 [4 to 5]

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- Stakeholder Advisory Group: To co-design an implementation strategy that targets critical components in the delivery of SCT or LCS services for patients who smoke.
  Convene a stakeholder advisory group (CHC providers, quality improvement specialists, community engagement staff, and specialty providers) to review the results of the literature review and quantitative analysis of deidentified data in order to select a set of implementation strategies from a menu of strategies to implement. The team will meet with the stakeholder advisory group five to six times for 0.5-1 hours each
  Qualitative Group Interviews: One time interview, 60-90 minutes
  Stakeholder advisory group: The team will meet with the stakeholder advisory group five to six times for 0.5-1 hours each
Arm/Group | Stakeholder Advisory Group
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/97/NCT05447897/Prot_SAP_000.pdf